CLINICAL TRIAL: NCT07008313
Title: Enhanced Recovery After Surgery Promotes the Rehabilitation of Patients With Acute Gastrointestinal Perforation, a Randomized Controlled Study
Brief Title: Enhanced Recovery After Surgery Promotes the Rehabilitation of Patients With Acute Gastrointestinal Perforation in Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Chunjie Liu, Professor, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HebMU 20180065
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Gastrointestinal Perforation; Enhanced Recovery After Surgery
Keywords: acute gastrointestinal perforation; enhanced recovery after surgery; perioperative period

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the enhanced recovery after surgery (ERAS) group (Experimental): Patients were rehabilitated using the ERAS concept.
  Interventions: Behavioral: The enhanced recovery after surgery
- the conventional surgical treatment (CST) group (Placebo Comparator): Traditional treatment methods.
  Interventions: Behavioral: Traditional treatment methods.

INTERVENTIONS:
Behavioral: The enhanced recovery after surgery — Enhanced recovery after surgery (ERAS) refers to a series of optimal management measures which are proved to be effective by evidence-based medical evidence in order to reduce patients' psychological and physiological traumatic stress reaction
  Arms: the enhanced recovery after surgery (ERAS) group
Behavioral: Traditional treatment methods. — Traditional treatment methods.
  Arms: the conventional surgical treatment (CST) group

SUMMARY:
The enhanced recovery after surgery(ERAS) has been gradually extended from its initial colorectal surgery to almost all surgical fields. However, there are few reports about the application value of ERAS in emergency surgery. The goal of this clinical trial is to evaluate the value of ERAS in the perioperative period of acute gastrointestinal perforation. All the patients will be treated by emergency operation. The changes of CRP, PA, PCT in Plasma 1 hour before operation and 1,3,7 days after operation, the operation time, the amount of bleeding during operation, the recovery time of intestinal function and the time of the first meal after operation,the incidence of postoperative complications, the degree of postoperative pain, the time of first out-of-bed activity, fatigue and mental status, quality of life, the length and the cost of hospital stay will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age≥14years old and ≤80 years old
* The initial diagnosis is acute gastrointestinal perforation

Exclusion Criteria:

* Patients with unconsciousness,or patients with past psychiatric history
* Patients with shock and/or severe organ failure
* Patients who are pregnant
* Patients with severe spinal deformity who are unable to receive epidural anesthesia

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
change of the c-reactive protein in plasma | 1, 3, and 7 days after surgery
change of the prealbumin in plasma | 1, 3, and 7 days after surgery
change of the procalcitonin in plasma | 1, 3, and 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China